CLINICAL TRIAL: NCT00698282
Title: A Randomised, Placebo-Controlled, Double-Blind, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Oral Doses of AZD1981 in Healthy Male Japanese and Caucasian Subjects
Brief Title: Single and Multiple Ascending Doses of AZD1981 in Japan
Acronym: JSAD/JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist, MD, Medical Science Director, R&D, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9831C00005
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
MeSH Terms: interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: AZD1981
- 2 (Experimental)
  Interventions: Drug: AZD1981
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1981 — Oral tablet, 250 mg single dose
  Arms: 1
Drug: AZD1981 — Suspension, 15, 75, 1000 and 2000 mg
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to study safety, tolerability and pharmacokinetics of AZD1981 in healthy Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese and Caucasian males

Exclusion Criteria:

* Other clinically relevant disease or disorders

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | All the time
Plasma drug concentration | Every hour

SECONDARY OUTCOMES:
Clinical chemistry | day 1 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hancox, Principal Investigator — Europe Chiltern International Ltd, Berkshire, UK
Locations (1):
- Research Site, Berkshire, United Kingdom